CLINICAL TRIAL: NCT05531630
Title: Xylitol Nasal Irrigations in the Treatment of Chronic Rhinosinusitis in Cystic Fibrosis Patients: a Randomized Crossover Trial
Brief Title: Xylitol vs Saline Nasal Irrigations in CF-CRS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S66364
Record Dates: First submitted 2022-08-19; First posted 2022-09-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: chronic rhinosinusitis; cystic fibrosis; nasal rinsing; xylitol; saline; nasal polyps
MeSH Terms: conditions — Disease; Cystic Fibrosis; Nasal Polyps

STUDY DESIGN:
Intervention Model Description: Patients will be asked to perform nasal irrigations with both Xylitol (treatment A) and saline (treatment B) once daily for six weeks, with a washout period of one week before the start of the treatment and one week between the two treatment periods. Washout periods are included to reduce the risk for a carryover effect. Patients will be randomized in two treatment arms: AB and BA. Patients in the AB arm will first receive Xylitol, followed by saline, and vice versa in the BA group.
Who Masked: Participant, Investigator
Masking Description: The study will be designed as a blinded trial, in which nor the investigator, nor the patient will know the sequence of the treatments (AB or BA). The patients will receive a box with sachets for treatment period 1 at the screening visit. The box will have a number from 1 to 76 and the sachets from both treatment groups will not contain any information regarding the content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB: Xylitol-Saline (Experimental): Patients in the AB arm will first receive Xylitol, followed by saline
  Interventions: Device: Nasal rinsing with saline 0.9%; Device: Nasal rinsing with Xylitol
- BA: Saline-Xylitol (Experimental): Patients in the BA arm will first receive saline, followed by Xylitol
  Interventions: Device: Nasal rinsing with saline 0.9%; Device: Nasal rinsing with Xylitol

INTERVENTIONS:
Device: Nasal rinsing with saline 0.9% — Nasal irrigations with saline (NaCl 0.9%) are considered golden standard in the treatment of chronic rhinosinusitis. Sachets consisting of mixtures for saline solutions, produced by DOS Medical®, consist of 1.875g sodium chloride and 0.625g sodium bicarbonate (figure 5). The content of the sachet has to be dissolved in 250mL heated water (lukewarm drinking water, max 37°C) in a NasoFree® nasal irrigator (Figure 4). Afterwards, the solution has to be mixed according to the instructions, the temperature has to be tested on the palm or forearm and afterwards, the product can be used. The patient will be asked to rinse their nose with the saline solution, once daily, for six weeks.
  The sachet with rinsing salt is considered to be a class I medical device and has a CE-label (CNK number 3309028).
Device: Nasal rinsing with Xylitol — Xylitol is a sugar-alcohol that is already implemented in the treatment of patients with (difficult-to-treat) chronic rhinosinusitis. Some (pilot) studies have already showed a positive effect in CRS patients without cystic fibrosis. Xylitol nasal rinsing salt, produced by DOS Medical®, is a mixture of 4g Xylitol, 1.875g sodium chloride, 0.625g sodium bicarbonate and 0,03g mint (Figure 3). The content of the sachet has to be dissolved in 250mL heated water (lukewarm drinking water, max 37°C) in a NasoFree® nasal irrigator (Figure 4). Afterwards, the solution has to be mixed according to the instructions, the temperature has to be tested on the palm or forearm and afterwards, the product can be used. The patient will be asked to rinse their nose with the Xylitol solution, once daily, for six weeks.
  The sachet with rinsing salt is considered to be a class I medical device, has a CE-label (CNK number 3309036) and is already commercially available in Belgium and The Netherlands.

SUMMARY:
Cystic fibrosis (CF) is the most common genetic disorder in Belgium, affecting 1 in 2850 children. A defect in the CFTR channel results in increased viscosity of extracellular secretions and decreased mucociliary clearance in the airways. As a result of this mechanism, chronic rhinosinusitis (CRS) occurs in nearly 100% of CF patients. CRS can lead to pronounced sinonasal complaints and can have a negative impact on the quality of life. In addition, several studies have shown that poor upper airway control has a negative impact on the lower airways. Unfortunately, treatment options are limited. Our previous study has shown that only 21% of patients have well-controlled CRS.

The aim of this single-center, randomized cross-over study is to compare the effect of nasal rinses with (XNI) and without (SNI) Xylitol in the treatment of CF-CRS. Xylitol is a sugar alcohol that is already used as an antibiofilm agent,eg in the prevention of caries. Previous pilot studies have already shown a beneficial effect of XNI in the treatment of non-CF CRS.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common genetic disorder in Belgium, affecting 1 in 2850 children. A defect in the CFTR channel results in increased viscosity of extracellular secretions and decreased mucociliary clearance in the airways. As a result of this mechanism, chronic rhinosinusitis (CRS) occurs in nearly 100% of CF patients. CRS can lead to pronounced sinonasal complaints and can have a negative impact on the quality of life of CF patients. In addition, several studies have shown that poor upper airway control has a negative impact on the lower airways. Unfortunately, treatment options are limited. Our previous study has shown that only 21% of patients have well-controlled CRS.

The aim of this study is to compare the effect of nasal rinses with (XNI) and without (SNI) Xylitol in the treatment of CF-CRS. Xylitol is a sugar alcohol that is already used as an antibiofilm agent, eg. in the prevention of caries.

Patients with cystic fibrosis, >18 years of age, who are known to have CRS with/without nasal polyps and who experience sinonasal symptoms in daily life, will be recruited (n=38). Patients with a visual analogue scale (VAS) score of >30/100 mm are included. Patients with a VAS <30 mm or patients who started <6 months ago with a CFTR modulator (eg Trikafta, Symkevi, Kalydeco) are excluded. After signing the ICF, patients are randomly allocated to a treatment arm "AB" or "BA". Patients in the study group 'AB' start, after a washout period of one week, with nasal rinses with Xylitol for six weeks. Afterwards, after another one week washout period, patients are asked to rinse the nose with standard saline nasal rinses without Xylitol for six weeks. Patients in the 'BA' group first start with standard nasal rinses, followed by Xylitol.

In total there are three planned study visits: a screening visit, a follow-up visit after the first treatment period and a follow-up visit after the second treatment period. During these visits, a nasal endoscopy (Lund-Kennedy and Modified Davos score) and smell tests (Sniffin' Sticks) are performed. In addition, the patients are asked to complete a questionnaire with VAS scores, the SNOT-22 score and the TRE score. Data is collected in a REDCAP database. Afterwards, the outcome parameters are statistically compared between the SNI and the XNI group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of cystic fibrosis > 18 years old
* Routine follow-up at UZ Leuven
* Patients with established diagnosis of chronic rhinosinusitis, with or without nasal polyps, and with a VAS-score of >30 out of 100 for at least one individual sinonasal symptom (nasal obstruction, rhinorrhea, postnasal drip, facial pain/pressure, reduced smell)
* Willing to participate in this study and compliant to the treatment

Exclusion Criteria:

* Patients <18 years old
* Start of CFTR gene-modulator less than 6 months prior to inclusion
* Not willing to participate in this trial or incompliant to the trial
* History of severe epistaxis (<6 months), requiring intervention by an ENT specialist
* History of hypersensitivity/allergic reaction/anaphylactic shock to one of the compounds of the sachets (NaCl, bicarbonate, mint, Xylitol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Visual analogue scale for total sinus symptom | 3 months
  questionnaire, scale from 0-100
Difference in SNOT-22 score | 3 months
  questionnaire, scale from 0-110
Difference in Thereapeutic response evaluation | 3 months
  questionnaire, scale from 1-5

SECONDARY OUTCOMES:
Difference in VAS for individual sinonasal symptoms | 3 months
  questionnaire, scale from 0-100
Difference in VAS for major sinus symptom | 3 months
  questionnaire, scale from 0-100
Difference in Lund-kennedy score | 3 months
  Endoscopy score (0-12)
Difference in Modified Davos score | 3 months
  Endoscopy score (0-8)
Difference in Olfactory function | 3 months
  Identification using Sniffin' sticks test, scale 0-16

CONTACTS AND LOCATIONS:
Overall Officials: Laura Van Gerven, MD, PhD, Principal Investigator — Department of Otorhinolaryngology, UZ Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No